CLINICAL TRIAL: NCT03772002
Title: Hepatitis C Surveillance With Linkage to Care of Patients From Non-infectious Departments in Tertiary Hospitals From Jiangsu, China
Brief Title: Hepatitis C Surveillance With Linkage to Care of Patients From Non-ID Departments in Jiangsu
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Chao Wu, Prof., The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IN-CN-987-5343
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCV screening (Experimental)
  Interventions: Diagnostic Test: HCV screening

INTERVENTIONS:
Diagnostic Test: HCV screening — HCV antibody and HCV RNA surveillance, anti-HCV treatment assessment

SUMMARY:
Due to the occult nature of hepatitis C virus (HCV), it is estimated that less than 5% of people with chronic hepatitis C (CHC) infection knowing their status. The major challenges are that awareness is lacking, reliable diagnostics and testing services are not sufficiently available, and laboratory capacity is weak. In the context of major tertiary hospitals, the well-functioning laboratories would ensure the high-quality HCV testing, which facilitate the identification of inpatients who are unaware of HCV infection. However, given the preliminary data, diagnostic rate of inpatients from non-infectious (non-ID) departments is disturbingly low. A recent study from a major hospital in Jilin province of China showed that 3.36% of inpatients were anti-HCV positive; however, HCV RNA confirmatory testing was not further performed in this study.

From the retrospective cohort in non-ID departments of a tertiary hospital of Jiangsu during 2016 to 2017, only 25.9% (71/273) of patients with anti-HCV antibody (Ab) further had HCV RNA confirmatory test, while 40% (29/71) were identified as CHC. The previous data indicates that insufficient anti-HCV Ab testing and insufficient follow-up of patients with positive anti-HCV Ab from non-ID departments. Indeed, compared to hospitals in Western countries, the infectious department in Chinese hospitals are relative independent from non-ID departments, meanwhile the knowledge of HCV infection is relatively lacking for non-ID physicians. Therefore, an appropriate clinical pathway for integration and linkage of non-ID department and ID departments for diagnosis and care delivery of CHC patients is urgently needed. The investigator aim to establish a feasible clinical pathway and consensus guideline to enhance HCV testing surveillance with linkage to care in non-ID departments. Moreover, the participants with anti-HCV Ab also will be enrolled in the HCV prospective cohort, in which the intervention and clinical outcome of hepatitis will be longitudinally monitored in the future study.

ELIGIBILITY:
Inclusion Criteria:

Retrospective cohort:

1. ≥ 18 years of age.
2. Inpatients from non-infectious department.
3. Documentation of laboratory test indicating positive HCV antibody.

Prospective cohort:

1. ≥ 18 years of age.
2. Inpatients from non-infectious departments.
3. Patients who meet the requirement of HCV antibody screening:

   1. patients with high risk possibility of HCV infection.
   2. patients who will have special or invasive medical operation.
   3. patients with unexplained abnormal liver biochemical laboratory results.

Exclusion Criteria:

Retrospective cohort: Duplicated subjects.

Prospective cohort：Inability or unwillingness to provide informed consent or abide by the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients in non-infectious departments who had positive HCV antibody testing but failed to get HCV RNA test. | 1 years
The percentage of HCV-RNA positivity among patients with the presence of anti-HCV antibody in non-infectious departments after Non-ID HCV screening. | 1 years
The percentage of HCV-RNA positivity linkage to care consensus guideline shaped. | 1 years

SECONDARY OUTCOMES:
The percentage of CHC patients linked to care in non-infectious departments. | 1 years
The treatment timeliness as embodied as time period from diagnosis to engagement to anti-HCV DAA treatment. | 1 years
The referral rate of identified HCV infected patients. | 1 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Third Hospital of Changzhou, Changzhou, Jiangsu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided